CLINICAL TRIAL: NCT03423316
Title: Stress-rest Calf Muscle Perfusion: a Functional Diagnostic Test for Peripheral Arterial Disease (PAD)
Brief Title: Functional MRI of the Lower Extremities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff L. Zhang, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P001781
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Controls (No Intervention)
- Age-Matched Controls (No Intervention): Subjects without PAD who have the same average age as the PAD patients
- PAD Patients (Experimental): Patients with PAD. Approximately 75% of PAD patients will be enrolled in the 12-week exercise therapy program.
  Interventions: Behavioral: Supervised exercise therapy

INTERVENTIONS:
Behavioral: Supervised exercise therapy — The therapy will be conducted three times each week for 12 weeks. Each session takes 1 hour, consisting of 5 minutes of warmup activities, 50 minutes of intermittent exercise, and 5 minutes of cool-down activities. Exercise consists of walking on a treadmill initiated at 2 mph and 0% grade, until claudication pain becomes moderately severe. After claudication pain subsides, the subject will restart the walk. At the end of the session, the total exercise duration will be recorded. After a patient is able to walk 8-10 minutes at the initial workload, the grade is increased by 1-2%, or the speed is increased by 0.5 mph as tolerated.
  Arms: PAD Patients

SUMMARY:
In this project, the investigators propose to use high-resolution magnetic resonance imaging (MRI) to measure blood perfusion in different groups of calf muscle. This imaging approach is standard of care for evaluation of coronary artery disease (CAD), and has never been successfully applied to PAD. Preliminary results show distinct patterns of muscle perfusion between healthy and PAD patients, and thus great promise of the technique. The investigators will first verify the reproducibility of the technique, and then compare the calf muscle perfusion measures in PAD patients against healthy age-matched controls. This comparison will test the feasibility of detecting functional abnormality in PAD patients. After the baseline scans, the PAD patients will opt to undergo a 12-week supervised exercise therapy, and then a post-therapy MRI scan. Comparison of the pre- and post-therapy measurements will indicate how the therapy improves the calf-muscle perfusion, and how this perfusion change correlates with increases in patient's walking ability.

The long term goals of this project are to develop an improved diagnostic test for patients with PAD to predict who will benefit from therapeutic intervention. The MRI perfusion studies of calf muscle can be performed in conjunction with routine peripheral MR angiography to assess the functional significance of vascular stenosis.

ELIGIBILITY:
Inclusion Criteria:

PAD patients with

* Intermittent claudication
* Ankle-brachial blood-pressure index (ABI) < 0.9

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Chronic pulmonary diseases
* Arthritis or other joint ailments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Stress-rest calf-muscle perfusion | Single visit (~90 minutes)
  Perfusion in the different calf muscle groups following exercises of low (rest) and high (stress) intensities
Perfusion changes following supervised exercise therapy | Before and after supervised exercise therapy (12 weeks)
  Change in stress-rest calf-muscle perfusion in PAD patients following the 12-week supervised exercise therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No